CLINICAL TRIAL: NCT04754503
Title: Survival and Quality of Life After Liver Transplantation in Patients Aged 65 and Over
Acronym: LT 65+
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A03063-36
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Patients Suitable for a Liver Transplant
Keywords: liver transplant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this non-interventional, single-center study is to assess survival and associated factors at 1 year in patients aged 65 and over who received liver transplantation

DETAILED DESCRIPTION:
The expected benefits of this study are to identify the preoperative risk factors of mortality from liver transplant failure in patients aged 65 and over (90-day mortality and 1 and 3-year survival) will allow better selection. candidates for this age group. In the current context of organ shortage, this study should make it possible to reduce the number of risky transplants and thus improve the allocation of grafts.Inclusion of patients who meet the inclusion criteria will be carried out during their hospitalization in the surgical department of the hepato-bilary center.

Included patients will receive a standardized geriatric assessment in addition to the usual assessment for a liver transplant.

The geriatric assessment will be carried out and conducted as follows: geriatric scores and quality of life questionnaires. Two geriatricians will perform the physical examination and blindly estimate each other's probability of survival at 90 days using a Likert scale.

Geriatricians will be blinded to hepatic data (reasons for transplantation). The consultation as well as the completion of the questionnaire will be carried out during the pre-transplantation assessment.

Survival and quality of life will be assessed at 3 and 12 months post-transplantaion.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for liver transplantation
* Having expressed non-oppostion to his participation in study and documented in his medical file
* With social coverage

Exclusion Criteria:

* Emergency transplant patients
* Patient already included in another study
* Patient under guardianship or curatorship
* Expressing his opposition to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients over 65 years of age who are candidates for a liver transplant at the participating center during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of survival and quality of life after liver transplantation according to the quality of life score | 12 Months

SECONDARY OUTCOMES:
Detecting depression in the elderly according the Geriatric Depression Scale (GDS) | 12 Months

OTHER OUTCOMES:
Assessment of commorbidity risk according Charlson score | At inclusion
Assessment of the degree of patient dependence according "Index of Independence in Activities of Daily Living" KATZ scale | 12 Months
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | 12 months
Assessment of quality of life according the SF-36 Health Status Questionnaire | 12 months
Assessment of the emotional, physical and financial burden on a caregiver according Zarit burden scale | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Duron Emmanuelle, MD PhD, Study Chair — Geriatric Department, Paul Brousse Hospital
Locations (1):
- Geriatric Department, Paul Brousse Hospital, Villejuif, Île-de-France Region, France